CLINICAL TRIAL: NCT04875845
Title: Comparison of Gastric Volume After 6-hour and 8-hour Fasting in Patient Scheduled for Elective Surgery
Status: Completed | Type: Observational
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Raden Besthadi Sukmono, Anesthesiologist, Regional Anesthesia Consultant, Assistant Professor, Indonesia University
Other Study IDs: GVES
Record Dates: First submitted 2021-04-21; First posted 2021-05-06 (Actual); Last update posted 2021-05-10 (Actual); Status verified 2021-05

CONDITIONS: Gastric Volume; Ultrasonography
Keywords: Gastric volume; preoperative fasting; ultrasonography.
MeSH Terms: interventions — Elective Surgical Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 6-hours fasting gastric volume: gastric volume measured after 6-hours fasting
  Interventions: Behavioral: Fasting for elective surgery
- 8-hours fasting gastric volume: gastric volume measured after 8-hours fasting
  Interventions: Behavioral: Fasting for elective surgery

INTERVENTIONS:
Behavioral: Fasting for elective surgery — 6-hours and 8-hours fasting before elective surgery

SUMMARY:
Preoperative fasting was a common practice to decrease perioperative aspiration risk. Duration of fasting was proportional to gastric volume. Short fasting duration may increase aspiration risk. However, prolonged perioperative fasting duration may lead to dehydration and hypoglycemia.

The objective of this study was to analyze gastric volume after 6-hour and 8-hour duration of fasting after consumption of solid meal on patients scheduled for elective surgery.

This was a cohort study recruiting 37 subjects from January to February 2019. Subjects were patients scheduled for elective non-digestive surgery in Cipto Mangunkusumo Hospital, Jakarta, Indonesia. Before fasting, all subjects consumed standard Cipto Mangunkusumo meal and was later assessed for gastric volume using ultrasound at 6 and 8 hour after meal was consumed.

DETAILED DESCRIPTION:
Background. Preoperative fasting was a common practice to decrease perioperative aspiration risk. Duration of fasting was proportional to gastric volume. Short fasting duration may increase aspiration risk. However, prolonged perioperative fasting duration may lead to dehydration and hypoglycemia. The protocols of 8 hours preoperative fasting was recommended by American Society of Anesthesiologist (ASA) after a full meal. The meal recognized by ASA to make this guidelines were Western diet that contains more fat. South East Asian (SEA) standard solid meal mainly contains rice and less protein and fats. We hypothesized 6-hours compared with 8-hours fasting was sufficient to provide ideal gastric volume for preoperative fasting after SEA standard solid meal. The objective of this study was to analyze gastric volume after 6-hour and 8-hour of fasting after consumption of SEA standard solid meal on patients scheduled for elective surgery.

Methods This was a cohort study recruiting 37 subjects from January to February 2019. Subjects were patients scheduled for elective non-digestive surgery in Cipto Mangunkusumo Hospital, Jakarta, Indonesia. Inclusion criteria were age between 18 to 60 years old, have no nutritional status disorder, and ASA physical status of 1 or 2. The exclusion criteria were patients with diabetes mellitus, pregnancy, abdominal distention, history of dyspepsia, and intestinal motility disturbances.

Subjects agreed to take part in the research, will be initial examined for obtaining demographic data: age, weight and height, type of surgery to be performed, and preoperative examinations. The subject will start 8 hours of fasting before the surgical planning time. Before fasting, the subjects were given Cipto Mangunkusumo Hospital food standardized nutritional levels. Subjects were given 1 hour to consume the food. Six hours after the standard meal is consumed, an ultrasound examination will be performed in the right lateral decubitus position to obtain ultrasound imaging of the antrum. After that, the subject continued fasting until 8 hours after meal and ultrasound examination was performed using the same technique to obtain images of ultrasound imaging of the antrum. Imaging pictures are taken at the time relaxation of the antrum, between two contractions. The results of this imaging are stored and assessments of antrum craniocaudal (CC) and anteroposterior (AP) diameters were performed by research assistants who don't know when the image was taken. These measurements were used to calculate Cross Sectional Area (CSA) using the formula of CSA=(π×CC×AP)/4. The Gastric Volume (GV) was then calculated with the formula GV=27.0+(14.6×CSA)-(1.28×age).

The primary data obtained was the result of repeated examinations. The analysis was adjusted using the Bonferonni correction factor. Categorical data was analyzed using the McNemar test. The results of data processing are displayed in tabular form. The gastric volume was grouped into sufficient and insufficient with a border value of 1.5ml/kg.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria were patients aged 18-60 years
* ASA 1-2 who would undergo non-digestive elective surgery in Cipto Mangunkusumo Hospital
* Body mass index between 20-30 kg/m2

Exclusion Criteria:

* patient who is not willing to enter the study
* patients with diabetes mellitus
* pregnancy
* abdominal distension
* intestinal motility disorders
* history of dyspepsia
* patients who do not receive the standard Cipto Mangunkusumo Hospital diet
* changes of the surgery schedule in which the patient is unable to do 8-hours fasting before surgery
* the patient who has an emergency in the perioperative period
* the patient was unable to consume the standard food provided

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: This was a cohort study for 37 subjects from January to February 2019. Subjects were patients scheduled for elective non-digestive surgery in Cipto Mangunkusumo Hospital
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Gastric Volume 6-hours | After 6-hours of preoperative fasting
  Gastric volume measured with ultrasound after 6-hours of preoperative fasting
Gastric Volume 8-hours | After 8-hours of preoperative fasting
  Gastric volume measured with ultrasound after 8-hours of preoperative fasting

CONTACTS AND LOCATIONS:
Overall Officials: Raden B Sukmono, Principal Investigator — Indonesia University
Locations (1):
- RSUPN Cipto Mangunkusumo, Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2019-06-13): https://cdn.clinicaltrials.gov/large-docs/45/NCT04875845/Prot_SAP_ICF_000.pdf